CLINICAL TRIAL: NCT00478387
Title: Study of the Immunogenicity of Killed Influenza Vaccine in Patients With Ovarian, Fallopian Tube, and Primary Peritoneal Cancer in Remission
Brief Title: Ovarian Cancer and Immune Response to Flu Vaccine
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 805443; UPCC 5806 (N01-A1-50024)
Record Dates: First submitted 2007-05-22; First posted 2007-05-24 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Ovarian Cancer
Keywords: Advanced Ovarian and Primary Peritoneal Cancer in Remission
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: The current season's trivalent killed influenza vaccine

SUMMARY:
The purpose of this study is to determine what the immune response is of ovarian cancer patients in remission, when they are given the flu vaccine. After receiving the flu vaccine, patients will have blood drawn 5 times in 12 months to study antibody response to the flu vaccine.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must have a histologic diagnosis of epithelial ovarian cancer or primary peritoneal carcinoma. Time from completion of chemotherapy will be no more than 6 months.
* If no clinical evidence of disease is present after diagnosis with Stage III or IV disease and completion of primary surgery and chemotherapy, or, if no clinical evidence of disease is present after completion of chemotherapy for a disease recurrence diagnosed after a progression-free interval of at least 2 years, for patients of any initial stage.

Exclusion Criteria:

* Prior malignancy (except basal cell or squamous cell skin cancer) within the past five years.
* Presence of active CNS disease.
* Active bacterial, viral or fungal infections.
* Chemotherapy, biologic therapy, or radiation therapy < 4 weeks prior to study entry.
* History of active autoimmunity or immunosuppression.
* Use of immunosuppressive drugs within 4 weeks prior to study entry. Patients may receive chemotherapy or other immunosuppressive medications at the discretion of their physician during the subsequent year after influenza vaccination without exclusion from the study.
* Patients with tumors of low malignant potential (borderline tumors) will not be eligible.
* Prior influenza vaccination with the current vaccine.
* History of serious sensitivity to eggs, or previous influenza vaccine.
* Pregnant of breastfeeding subjects.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To gather preliminary information regarding immune response following influenza vaccination via measurement of antibody in subjects with advanced ovarian and primary peritoneal cancer in remission..
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2006-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina S Chu, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Department of Obstetrics and Gynecology, Division of GYN Oncology, Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States